CLINICAL TRIAL: NCT06979284
Title: Intravascular Ultrasound for Peripheral Artery Disease Revascularization: The CLARITY Randomized Controlled Trial
Brief Title: Intravascular Ultrasound for Peripheral Artery Disease Revascularization
Acronym: CLARITY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5251
Record Dates: First submitted 2025-05-02; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-04

CONDITIONS: Peripheral Arterial Disease(PAD); Chronic Limb Threatening Ischemia; Intravascular Ultrasound; Major Adverse Limb Events; Restenosis
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Intervention Model Description: Multicenter, international, prospective, randomized, open, blinded endpoint (PROBE) parallel trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravascular Ultrasound - guided strategy (Active Comparator): Percutaneous revascularization will be performed using intravascular ultrasound.
  Interventions: Procedure: IVUS-guided strategy
- Angiography - guided strategy (No Intervention): A standard-of-care percutaneous revascularization will be performed without using intravascular ultrasound.

INTERVENTIONS:
Procedure: IVUS-guided strategy — Percutaneous revascularization will be performed using intravascular ultrasound. The operators will follow instructions to modify arteries hardened by calcium and use IVUS to optimize the equipment (balloon and stents) used to unblock the artery.
  Arms: Intravascular Ultrasound - guided strategy

SUMMARY:
The purpose of this study is to determine if IVUS use, as compared to angiography alone, prevent major adverse limb events (MALE) or binary restenosis (a greater than 50% re-narrowing of the treated artery) in adult patients who have CLTI and are undergoing percutaneous revascularization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with lower extremity PAD manifesting as CLTI:

   a. CLTI is defined as ischemic rest foot pain, nonhealing wounds, or gangrene present for at least two weeks and that is attributable to objectively proven arterial occlusive disease, compatible with Rutherford class 4, 5 or 6, with the following supporting hemodynamic criteria1: i. For ischemic rest pain (Rutherford category 4): Ankle systolic pressure < 40mmHg, toe pressure < 30mmHg, or flat-line transtarsal pulse volume recording, OR ii. For tissue loss (Rutherford category 5, 6): Ankle systolic pressure < 60 mmHg, toe pressure of < 40mmHg, or flat-line transtarsal volume recording, AND
2. Scheduled to undergo percutaneous revascularization, AND
3. Informed consent
4. Imaging evidence of an obstructive or occluded lesion (> 70%) in the infraiguinal circulation (e.g. femoral, popliteal, or infrapopliteal circulation) using angiography, ultrasound, computed tomography, or magnetic resonance imaging.
5. An infrapopliteal lesion must be located in the proximal 2/3 of native infrapopliteal vessels, with a vessel diameter of > 2.5mm by investigator visual assessment.
6. The distal margin of the most distal target lesion must be located > 10 cm proximal to the proximal margin on the ankle mortise. The vessel segment distal to the most distal target lesion must be patent all the way to the ankle, with no obstructive lesion (>50% stenosis).

Exclusion Criteria:

1. The presence of anatomic or comorbid conditions or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the potential participant's ability to participate in the trial or to comply with the follow-up requirements.
2. The presence of any medical conditions precluding percutaneous revascularization
3. The subject has previously had or requires surgical revascularization involving the vessel containing the target lesion of the ipsilateral extremity.
4. The subject is bedridden or unable to walk (with assistance is acceptable).
5. Life expectancy < 12 months
6. Age < 18 years
7. Active vasculitis, Buerger's disease, or acute limb-threatening ischemia
8. Planned above-ankle amputation of the index limb within four weeks of the index procedure.
9. Obstructive supra-inguinal "inflow" (>70% stenosis) which is not planned to be treated during index procedure or within 30 days of the index procedure.
10. The subject has had any amputation to the ipsilateral extremity other than the toe or forefoot, or the subject has had a major amputation to the contralateral extremity < 1 year before the index procedure and is not independently walking.
11. Extensive tissue loss that is salvageable only with complex foot reconstruction or non-traditional trans metatarsal amputations.

    1. Osteomyelitis that extends proximal to the metatarsal heads
    2. Gangrene involving the plantar skin of the forefoot, midfoot or heel
    3. Deep ulcer or large shallow ulcer (> 3 cm) involving the plantar skin of the f forefoot, midfoot, or heel
    4. Full-thickness heel ulcer
    5. Any wound with calcaneal bone involvement
    6. Wounds that would require flap coverage or complex wound management for large soft tissue defect
    7. Full-thickness wounds on the dorsum of the foot with exposed tendon or bone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 772 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2030-07 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Time-to-first occurrence of MALE | From date of randomization until the date of first unplanned above ankle amputation of the index limb, clinically driven target lesion revascularization or target-lesion binary restenosis, assessed up to a maximum of 5 years.
  Defined as unplanned above ankle amputation of the index limb or clinically driven target lesion revascularization, or target-lesion binary restenosis, defined as > 50% stenosis on imaging throughout follow-up.

SECONDARY OUTCOMES:
The composite of all-cause mortality, MALE, or target-lesion binary restenosis | From date of randomization until the date of death, MALE, or target lesion binary restenosis, assessed up to a maximum of 5 years.
MALE | From date of randomization, assessed up to a maximum of 5 years.
All-cause mortality | From date of randomization, assessed up to a maximum of 5 years.
Unplanned above-ankle amputation of the index limb | From date of randomization, assessed up to a maximum of 5 years.
Clinically-driven target lesion revascularization | From date of randomization, assessed up to a maximum of 5 years.
Target lesion binary restenosis | From date of randomization, assessed up to a maximum of 5 years.
Unplanned minor amputation of the index limb | From date of randomization, assessed up to a maximum of 5 years.
Wound healing status of the index limb based on the Wound, Ischemia, Foot Infection (WIFI) scale throughout follow-up | From date of randomization, assessed up to a maximum of 5 years.
  The WIFI assessment refers to the Wound, Ischemia, and Foot Infection (WIFI) classification system. This system is used to standardize the measurement of wound healing, particularly in patients with peripheral artery disease (PAD). It is not a questionnaire but rather a classification method that helps in assessing the severity of wounds, the degree of ischemia (restricted blood supply), and the presence of foot infections. Wound, Ischemia and foot infection are all graded on a scale of 0-3, with higher grades indicating more severe conditions.
Change in the Walking Impairment Questionnaire (WIQ) score throughout follow-up | From date of randomization, assessed up to a maximum of 5 years.
  The Walking Impairment Questionnaire (WIQ) is a tool designed to measure walking ability in patients with Peripheral Arterial Disease (PAD). It assesses the impact of PAD on walking distance, walking speed, and the ability to climb stairs. The WIQ is particularly useful for evaluating the severity of walking impairment and the effectiveness of interventions aimed at improving walking ability in these patients. The WIQ includes several categories, each scored on a scale from 0 to 100, with higher scores indicating better walking ability.
  Each category score is calculated based on the patient's self-reported ability to perform these activities. The scores are then used to provide an overall assessment of the patient's walking impairment.
Change in the Vascular Quality of Life Questionnaire-6 (VascQol-6) score throughout follow-up | From date of randomization, assessed up to a maximum of 5 years.
  The VascuQoL-6 questionnaire is a health-related quality of life (QoL) assessment tool specifically designed for patients with peripheral arterial disease (PAD). It is used in clinical practice and vascular registries to evaluate the impact of PAD on patients' quality of life.
  Scale Determination The VasQol-6 consists of six questions, each scored on a scale from 1 to 4. The scores for each question are summed to generate a total Quality of Life score. A higher total score indicates a better health status.
  Score 1: Indicates the worst health status. Score 4: Indicates the best health status.